CLINICAL TRIAL: NCT00002938
Title: The Role of Salvage Prostatectomy for Radiation Failure in Prostate Carcinoma: A Phase II Trial
Brief Title: Surgery in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-9687; U10CA031946 (NIH); CALGB-9687; CDR0000065381 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Other): Salvage prostatectomy
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Procedure: conventional surgery — Salvage prostatectomy

SUMMARY:
RATIONALE: Prostatectomy may be an effective treatment for prostate cancer that has not responded to radiation therapy.

PURPOSE: This phase II trial is studying how well prostatectomy works in treating patients with recurrent or persistent prostate cancer that has not responded to radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the characteristics of failure-free survival, disease-free survival, overall survival, surgical morbidity and mortality, and quality of life of patients treated with salvage prostatectomy for the recurrence of persistent disease after treatment with prior radiotherapy for localized prostate cancer.
* Develop expertise in the use of salvage prostatectomy prior to a possible phase III trial of salvage prostatectomy in this population versus a control arm such as hormonal therapy or cryotherapy.
* Determine the quality of life measures in these patients.
* Determine the preliminary data on the quality of life of patients undergoing salvage radical prostatectomy and use the data to design a phase III study.
* Determine the histologic and morphometric characterization of the carcinoma.

OUTLINE: Patients undergo modified bilateral pelvic lymph node dissection.

Patients with negative nodes undergo salvage prostatectomy via either retropubic or perineal approach. Patients with positive nodes may undergo radical prostatectomy at the discretion of the investigator.

Postoperative hormonal therapy may be given at time of symptomatic disease progression or a newly positive bone scan, or for a consistently rising prostate-specific antigen. Adjuvant hormonal therapy is also allowed.

Quality of life is assessed prior to surgery and at 3, 6, 12, 18, and 24 months after surgery.

Patients are followed at least every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent or persistent prostate cancer
* Prostate-specific antigen (PSA) no greater than 20 ng/mL
* Must have been previously treated with at least 60 cGy of external beam radiotherapy or brachytherapy for clinical stages T1-2NXM0 with PSA no greater than 30 ng/mL
* No metastatic disease at time of biopsy

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* CALGB (Zubrod) 0-1

Life expectancy:

* At least 5-10 years

Other:

* No other "currently Temporarily closed" malignancy except nonmelanoma skin cancer

  * Patients are not considered to have a "currently Temporarily closed" malignancy if they have completed therapy and are considered to be at less than 30% risk of relapse

PRIOR CONCURRENT THERAPY:

Endocrine therapy:

* At least 3 months since prior adjuvant hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 18 months since prior external beam or interstitial radiotherapy

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 1997-05; Primary Completion 2005-02 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Survival characteristics | pre treatment; q 3 mon for 2 years, then q 6 mon for 2 yrs, then q year

SECONDARY OUTCOMES:
QOL assessment | pre treatment; 3, 6, 12, 18, and 24 mon post treatment
  Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gary D. Steinberg, MD, Study Chair — University of Chicago
Locations (61):
- United States (61):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Comprehensive Cancer Center at Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Miriam Hospital at Lifespan, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Sokoloff MH, Halabi S, Sanford B, et al.: Management of recurrent prostate cancer after radiotherapy: preliminary results of CALGB 9687, a contemporary salvage prostatectomy series. [Abstract] American Society of Clinical Oncology 2005 Prostate Cancer Symposium, 17-19 February 2005, Orlando, Florida. A-166, 2005.